CLINICAL TRIAL: NCT07340242
Title: Dentoskeletal Effects of CAD/CAM 3D-Printed Fixed Twin Block Versus MARA Appliances in the Management of Skeletal Class II Due to Mandibular Deficiency in Preadolescence: A Randomized Controlled Trial
Brief Title: Dentoskeletal Effects of 3D-Printed Fixed Twin Block Versus MARA Appliances in Management of Skeletal Class II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Yasmin Ghaly, Assistant Lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDP.25.03.5
Record Dates: First submitted 2025-11-21; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Class II Malocclusion; Mandibular Deficiency
MeSH Terms: conditions — Overbite; Micrognathism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group, who will be the untreated group. (No Intervention)
- . MARA group, who will undergo MARA appliance (Active Comparator)
  Interventions: Device: MARA appliance
- Fixed twin block group, who will undergo fixed twin block appliance (Active Comparator)
  Interventions: Device: fixed twin block

INTERVENTIONS:
Device: MARA appliance — CAD/CAM 3D printed mandibular anterior repositioning appliance
  Arms: . MARA group, who will undergo MARA appliance
Device: fixed twin block — CAD/CAM 3D printed fixed twin block
  Arms: Fixed twin block group, who will undergo fixed twin block appliance

SUMMARY:
Objective: to evaluate the dentoskeletal effects of CAD/CAM 3D-Printed fixed twin block versus MARA appliances in the management of skeletal class II due to Mandibular Deficiency in Preadolescence Class II malocclusion is considered one of the most commonly observed problems among orthodontic patients, representing around one-third of the patients seeking orthodontic treatment reflecting a significant economic impact. Various removable and fixed functional appliances are commonly used to stimulate mandibular growth. Fixed Twin-block appliance has advantages compared with removable Twin-block and Herbst appliances. The mandibular anterior repositioning appliance is referred to as M.A.R.A. appliance.

Materials and method: The study design is a randomized controlled trial in which the control group and intervention groups will be assessed as parallel groups with a 1:1:1 allocation ratio. Sixty subjects will be enrolled in this research. They will be divided equally into three groups: untreated control, MARA group and Twin block group

ELIGIBILITY:
Inclusion Criteria:

1. Skeletal Class II malocclusion due to mandibular retrusion.
2. Overjet ≥ 6.0 mm.
3. Normal or low-angle growth pattern.
4. Minimum crowding in the mandibular arch.
5. Undergoing circumpubertal phase of skeletal development (CVMI 2, 3, and 4)

Exclusion Criteria:

1. Clinical signs and symptoms of temporomandibular disorder.
2. Systemic disease affecting bone and general growth.
3. Previous orthodontic treatment
4. Cleft lip or palate.
5. Congenital craniofacial deformity.
6. Abnormal oral habits.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-04-27 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-04-27 (Estimated)

PRIMARY OUTCOMES:
Linear Skeletal changes of the maxilla and mandible using cephalometric measurements | From date of randomization until the date of first documented acceptable correction assessed up to 6 months
  linear (mm) measurement
Angular skeletal changes of the maxilla and mandible using cephalometric measurements | From date of randomization until the date of first documented acceptable correction assessed up to 6 months
  angular (°) measurement
Linear dental changes of the maxilla and mandible using cephalometric measurements | From date of randomization until the date of first documented acceptable correction assessed up to 6 months
  linear (mm) measurement
Angular dental changes of the maxilla and mandible using cephalometric measurements | From date of randomization until the date of first documented acceptable correction assessed up to 6 months
  angular (°) measurement
Linear soft tissue changes of the maxilla and mandible using cephalometric measurements | From date of randomization until the date of first documented acceptable correction assessed up to 6 months
  linear (mm) measurement
Angular soft tissue changes of the maxilla and mandible using cephalometric measurements | From date of randomization until the date of first documented acceptable correction assessed up to 6 months
  angular (°) measurement

SECONDARY OUTCOMES:
Oral health quality of life questionnaire | From date of randomization until the date of first documented acceptable correction assessed up to 6 months
  The questionnaire (COHIP-SF-AR) will be given to the participants once informed consent is obtained at 5-time points: before treatment, 1 week, 1 month, 3 months, and 6 months after wearing functional appliances.
Incidence of breakages and harms reported during routine or emergency visits in both groups | From date of randomization until the date of first documented acceptable correction assessed up to 6 months
  Details of complications in both groups, including breakages and harms reported during routine or emergency visits, will be registered and categorized according to their nature and severity using a previously published classification system
Arch perimeter and depth measurement from digital model analysis | From date of randomization until the date of first documented acceptable correction assessed up to 6 months
  linear (mm) measurement
Maxillary inter-canine width from digital model analysis | From date of randomization until the date of first documented acceptable correction assessed up to 6 months
  linear (mm) measurement
Maxillary inter-first molar width from digital model analysis | From date of randomization until the date of first documented acceptable correction assessed up to 6 months
  linear (mm)measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided